CLINICAL TRIAL: NCT00973414
Title: Fluid Management for Cesarean Section Undergoing Combined Spinal Epidural Anesthesia (CSEA)
Brief Title: Fluid Management for Cesarean Section III
Acronym: FMCS-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NJMU-09053MZ
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Cesarean Section
Keywords: Combined epidural spinal anesthesia; Fluid therapy
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prior crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) was given before CSEA
  Interventions: Drug: Ringer's Lactate
- Posterior crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) was given after CSEA
  Interventions: Drug: Ringer's Lactate
- Prior colloid (Active Comparator): Colloid (6% hydroxyethyl starch) was given before CSEA
  Interventions: Drug: Six percent hydroxyethyl starch
- Posterior colloid (Active Comparator): Colloid (6% hydroxyethyl starch) was given after CSEA
  Interventions: Drug: Six percent hydroxyethyl starch

INTERVENTIONS:
Drug: Ringer's Lactate — Ringer's Lactate 8 ml/kg was given intravenously before or after CSEA in cesarean section
  Other Names: Lactated Ringer's solution
  Arms: Posterior crystalloid; Prior crystalloid
Drug: Six percent hydroxyethyl starch — Hydroxyethyl starch (6%) was given before or after CSEA in cesarean section
  Other Names: HES/HAES
  Arms: Posterior colloid; Prior colloid

SUMMARY:
Regional anesthesia, including epidural, spinal and combined epidural spinal anesthesia (CSEA), is a pivotal part in modern anesthesiology. Previously, the investigators found that epidural and spinal anesthesia during cesarean section possesses different responsiveness to fluid (including crystalloid and colloid) management given prior or posterior to anesthesia. Although CSEA is also widely used as an alternative of single epidural or spinal anesthesia for its combined effect of fast onset of anesthesia of spinal anesthesia and the property of duration of epidural catheterization, the fluid resuscitation during CSEA is still unknown. The investigators hypothesized that fluid management during CSEA would produce different effect on hemodynamics in cesarean section compared with epidural and spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 yr
* First time of delivery
* ASA status I-II
* No premature
* No genetic and infectious diseases
* Chinese

Exclusion Criteria:

* < 21 yr
* > 40 yr
* Subjects with cardiac and pulmonary disorders
* Dislocation of placenta
* Pregnant hypertension
* Allergy to local anesthetics
* Unwilling to cooperation
* Need intraoperative administration of vascular active agents
* With significant delivery side effects

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 850 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Rate of hypotension | Anesthesia begin (0 min) to 120 min after anesthesia

SECONDARY OUTCOMES:
Recurrence of hypotension after ephedrine or phenylephrine | Anesthesia begin (0 min) to 120 min after anesthesia
Consumption of ephedrine and phenylephrine | Anesthesia begin (0 min) to 120 min after anesthesia
Total volume of colloid or crystalloid | Fifteen minutes before anesthesia to 120 min after anesthesia
One-min and 5-min Apgar scores | The first and fifth minute after cesarean successful delivery
Oxygen saturation during hypotension | Anesthesia begin (0 min) to 120 min after anesthesia
Duration of hypotension | Anesthesia begin (0 min) to 120 min after anesthesia
Low umbilical cord pH (artery < 7.20) | At the time of successful delivery (0 min)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- The Affiliated Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China